CLINICAL TRIAL: NCT01258985
Title: Tai Chi and Physical Therapy for Knee Osteoarthritis
Acronym: TCPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01AT005521-01A1 (NIH); R01AT005521 (NIH); UL1TR000073 (NIH); UL1TR001064 (NIH)
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Results first posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-06

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Knee osteoarthritis; osteoarthritis; Knee pain; Tai Chi; Physical Therapy; mind-body exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Tai Ji; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tai Chi (Active Comparator): 12 weeks of Tai Chi classes
  Interventions: Behavioral: Tai Chi
- Physical Therapy (Active Comparator): 6 weeks of individualized Physical Therapy followed by 6 weeks of Supervised Home Exercise
  Interventions: Behavioral: Physical Therapy

INTERVENTIONS:
Behavioral: Tai Chi — 12 weeks of Tai Chi
  Arms: Tai Chi
Behavioral: Physical Therapy — 6 weeks of individualized Physical Therapy followed by 6 weeks of supervised Home Exercise
  Arms: Physical Therapy

SUMMARY:
We will conduct a large randomized controlled trial comparing the effectiveness and cost-effectiveness of Tai Chi mind-body exercise and standard-of-care Physical Therapy for Knee Osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) causes pain and long-term disability, and the public health impact will increase as the population ages. In addition to inconsistent effectiveness, current treatments such as nonsteroidal anti-inflammatory drugs, knee replacement, and physical therapy may be expensive, result in serious adverse effects, reduce physical function, and fail to improve mental well-being. Finding effective treatments to maintain function and quality of life in OA patients is one of the national priorities identified this year by the Institute of Medicine.

We propose to conduct the first comparative effectiveness and cost-effectiveness trial of Tai Chi vs. physical therapy (PT) in a large symptomatic Knee OA population. A single-blind, randomized, controlled trial of Tai Chi vs. Physical Therapy will be conducted in 180 patients who meet the American College of Rheumatology criteria for Knee OA. Patients will be randomized to 12 weeks of treatment with Tai Chi (2x/week) or Standard Physical Therapy (2x/week for 6 weeks, followed by 6 weeks of rigorous supervised home exercise) with 24 and 52 week follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years and older
* American College of Rheumatology criteria for symptomatic Knee OA: Pain on more than half the days of the past month during at least one of the following activities: walking, going up or down stairs, standing upright, or lying in bed at night;101 radiographic evidence of grade I-III tibiofemoral or patellofemoral OA: defined as the presence of osteophytes in the tibiofemoral compartment and /or the patellofemoral compartment, as assessed on standing anterior/posterior and lateral views101
* WOMAC pain subscale score >= 40 (visual analog version) on at least 1 of 5 questions (range 0 to 100 each)
* Clinical examination confirming knee pain or discomfort or instability referable to the knee joint
* Physically able to participate in both the Tai Chi and Standard PT programs
* Willing to undergo testing and intervention procedures and 1.willing to abstain from Tai Chi until completion of the program, if randomized to Standard PT regimen. 2. willing to abstain from Standard PT regimen until completion of the program, if randomized to Tai Chi

Exclusion Criteria:

* Prior experience with physical therapy, Tai Chi or other similar types of Complementary and Alternative Medicine in the past 1 year such as Qi gong and yoga since these share some of the principles of Tai Chi.
* Serious medical conditions limiting the ability and safety to participate in either the Tai Chi or Standard PT regimen programs as determined by primary care physicians; these include dementia, neurological disease, symptomatic heart or vascular disease (angina, peripheral vascular disease, congestive heart failure), severe hypertension, recent stroke, severe insulin-dependent diabetes mellitus, psychiatric disease, renal disease, liver disease, active cancer and anemia
* Any intra-articular steroid injections in the previous 3 months or reconstructive surgery on the affected knee
* Any intra-articular Synvisc or Hyalgan injections in the previous 6 months
* Inability to pass the Mini-Mental Status examination (with a score below 24)102
* Inability to walk without a cane or other assistive device 100% of the time during the baseline assessments
* Enrollment in any other clinical trial within the last 30 days
* Plan to permanently relocate from the region during the trial period
* Positive pregnancy test or planning pregnancy within the study period
* Not English-Speaking

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2011-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chenchen Wang, MD, MSc, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available upon request.

REFERENCES:
- [Background] Wang C, Collet JP, Lau J. The effect of Tai Chi on health outcomes in patients with chronic conditions: a systematic review. Arch Intern Med. 2004 Mar 8;164(5):493-501. doi: 10.1001/archinte.164.5.493. PMID 15006825
- [Background] Wang C, Roubenoff R, Lau J, Kalish R, Schmid CH, Tighiouart H, Rones R, Hibberd PL. Effect of Tai Chi in adults with rheumatoid arthritis. Rheumatology (Oxford). 2005 May;44(5):685-7. doi: 10.1093/rheumatology/keh572. Epub 2005 Mar 1. No abstract available. PMID 15741197
- [Background] Wang C. Tai Chi improves pain and functional status in adults with rheumatoid arthritis: results of a pilot single-blinded randomized controlled trial. Med Sport Sci. 2008;52:218-229. doi: 10.1159/000134302. PMID 18487901
- [Background] Wang C, Schmid CH, Rones R, Kalish R, Yinh J, Goldenberg DL, Lee Y, McAlindon T. A randomized trial of tai chi for fibromyalgia. N Engl J Med. 2010 Aug 19;363(8):743-54. doi: 10.1056/NEJMoa0912611. PMID 20818876
- [Background] Wang C, Schmid CH, Hibberd PL, Kalish R, Roubenoff R, Rones R, McAlindon T. Tai Chi is effective in treating knee osteoarthritis: a randomized controlled trial. Arthritis Rheum. 2009 Nov 15;61(11):1545-53. doi: 10.1002/art.24832. PMID 19877092
- [Background] Wang C, Schmid CH, Hibberd PL, Kalish R, Roubenoff R, Rones R, Okparavero A, McAlindon T. Tai Chi for treating knee osteoarthritis: designing a long-term follow up randomized controlled trial. BMC Musculoskelet Disord. 2008 Jul 29;9:108. doi: 10.1186/1471-2474-9-108. PMID 18664276
- [Background] Reid KF, Price LL, Harvey WF, Driban JB, Hau C, Fielding RA, Wang C. Muscle Power Is an Independent Determinant of Pain and Quality of Life in Knee Osteoarthritis. Arthritis Rheumatol. 2015 Dec;67(12):3166-73. doi: 10.1002/art.39336. PMID 26315282
- [Derived] Lee AC, Harvey WF, Price LL, Han X, Driban JB, Iversen MD, Desai SA, Knopp HE, Wang C. Dose-Response Effects of Tai Chi and Physical Therapy Exercise Interventions in Symptomatic Knee Osteoarthritis. PM R. 2018 Jul;10(7):712-723. doi: 10.1016/j.pmrj.2018.01.003. Epub 2018 Jan 31. PMID 29407226
- [Derived] Lee AC, Harvey WF, Price LL, Han X, Driban JB, Wong JB, Chung M, McAlindon TE, Wang C. Mindfulness Is Associated With Treatment Response From Nonpharmacologic Exercise Interventions in Knee Osteoarthritis. Arch Phys Med Rehabil. 2017 Nov;98(11):2265-2273.e1. doi: 10.1016/j.apmr.2017.04.014. Epub 2017 May 12. PMID 28506776
- [Derived] Lee AC, Driban JB, Price LL, Harvey WF, Rodday AM, Wang C. Responsiveness and Minimally Important Differences for 4 Patient-Reported Outcomes Measurement Information System Short Forms: Physical Function, Pain Interference, Depression, and Anxiety in Knee Osteoarthritis. J Pain. 2017 Sep;18(9):1096-1110. doi: 10.1016/j.jpain.2017.05.001. Epub 2017 May 10. PMID 28501708
- [Derived] Wang C, Schmid CH, Iversen MD, Harvey WF, Fielding RA, Driban JB, Price LL, Wong JB, Reid KF, Rones R, McAlindon T. Comparative Effectiveness of Tai Chi Versus Physical Therapy for Knee Osteoarthritis: A Randomized Trial. Ann Intern Med. 2016 Jul 19;165(2):77-86. doi: 10.7326/M15-2143. Epub 2016 May 17. PMID 27183035
- [Derived] Driban JB, Morgan N, Price LL, Cook KF, Wang C. Patient-Reported Outcomes Measurement Information System (PROMIS) instruments among individuals with symptomatic knee osteoarthritis: a cross-sectional study of floor/ceiling effects and construct validity. BMC Musculoskelet Disord. 2015 Sep 14;16:253. doi: 10.1186/s12891-015-0715-y. PMID 26369412
- [Derived] Wang C, Iversen MD, McAlindon T, Harvey WF, Wong JB, Fielding RA, Driban JB, Price LL, Rones R, Gamache T, Schmid CH. Assessing the comparative effectiveness of Tai Chi versus physical therapy for knee osteoarthritis: design and rationale for a randomized trial. BMC Complement Altern Med. 2014 Sep 8;14:333. doi: 10.1186/1472-6882-14-333. PMID 25199526

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tai Chi | Physical Therapy
Started | 106 | 98
Completed | 106 | 98
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tai Chi | Physical Therapy | Total
Number analyzed (Participants) | 106 | 98 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (10.5) | 60.1 (10.5) | 60.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 68 | 143
  Male | 31 | 30 | 61
Race/Ethnicity, Customized [Number; unit: participants]
  White | 54 | 54 | 108
  Black | 41 | 31 | 72
  Asian | 4 | 2 | 6
  Other | 7 | 11 | 18
Region of Enrollment [Number; unit: participants]
  United States | 106 | 98 | 204

OUTCOME MEASURES:

1. Primary Outcome: Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC)Pain Subscale From Baseline to 12 Weeks
Description: The WOMAC (version: Visual Analog Scale 3.1) is a validated, self-administered, visual analogue scale specifically designed to evaluate knee and hip osteoarthritis. It has three subscales that are analyzed separately: pain (score range, 0-500), stiffness (0-200), and function (0-1700), with higher scores indicating more severe disease.
Time Frame: From Week 0 to Week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi | Physical Therapy
Number analyzed (Participants) | 106 | 98
units on a scale | -167.2 [-190.4 to -144.9] | -143 [-167.4 to -118.6]

2. Secondary Outcome: Change in Medical Outcomes Short Form-36 PCS
Description: The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) Physical Component Score (PCS) is the summary score for the physical quality-of-life components (range, 0 to 100, with higher scores indicating better health status)
Time Frame: From Week 0, to Week 12, or to week 24, or to week 52
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi | Physical Therapy
Number analyzed (Participants) | 106 | 98
units on a scale
  week 12 | 6.3 [4.6 to 7.9] | 3.1 [1.4 to 4.8]
  24 weeks | 7.1 [5.1 to 9.0] | 3.4 [1.4 to 5.5]
  52 weeks | 6.3 [4.4 to 8.3] | 4.3 [2.3 to 6.4]

3. Secondary Outcome: Change in 6 Minute Walk
Description: The 6 minute Walk Test is a measure of functional exercise capacity. Participants are asked to walk as far as possible within a six-minute period, and the distance covered at the end is noted and recorded.
Time Frame: From Week 0, to Week 12, or to week 24, or to week 52
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Tai Chi | Physical Therapy
Number analyzed (Participants) | 106 | 98
meters
  Week 12 | 28.6 [17.9 to 39.2] | 26.1 [14.9 to 37.4]
  Week 24 | 28.9 [16.6 to 41.2] | 24.5 [11.5 to 37.5]
  Week 52 | 27.1 [12.2 to 42.0] | 22.8 [7.0 to 38.6]

4. Secondary Outcome: Change in 20 Meter Walk Test
Description: the 20-meter walk test is a performance measurement of walking ability (measured as the total number of seconds it takes to walk 20 meters); lower scores indicate improved walking ability
Time Frame: From Week 0, to Week 12, or to week 24, or to week 52
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Tai Chi | Physical Therapy
Number analyzed (Participants) | 106 | 98
seconds
  12 weeks | -1.6 [-2.4 to -0.8] | -1.1 [-2.0 to -0.2]
  24 weeks | -2.4 [-3.4 to -1.3] | -1.2 [-2.2 to -0.1]
  52 weeks | -2.4 [-3.5 to -1.4] | -1.0 [-2.1 to 0.2]

5. Secondary Outcome: Change in Patient Global VAS
Description: Patients' global assessment score (Patient Global VAS) was assessed separately by the participant, who was unaware of the group assignment, with the use of a visual-analogue scale (VAS) (range, 0 to 10,with higher scores indicating greater pain).
Time Frame: From Week 0, to Week 12, or to week 24, or to week 52
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi | Physical Therapy
Number analyzed (Participants) | 106 | 98
units on a scale
  12 weeks | -0.3 [-0.3 to -0.2] | -0.2 [-0.3 to -0.2]
  24 weeks | -2.4 [-2.93 to -1.88] | -1.73 [-2.29 to -1.17]
  52 weeks | -1.84 [-2.48 to -1.21] | -1.31 [-1.96 to -0.66]

6. Secondary Outcome: Change in Beck II Depression Inventory
Description: Beck II Depression Inventory (BDI), second edition, is a 21-question, validated, self-report instrument that measures the severity of depressive symptoms. Total scores range from 0-63, and higher scores reflect greater depressive symptoms. BDI scores ranging from 0-13 represent minimal depressive symptoms; scores from 14-19 are mild; scores from 20-28 are moderate; and scores from 29-63 represent severe depressive symptoms.
Time Frame: From Week 0, to Week 12, or to week 24, or to week 52
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi | Physical Therapy
Number analyzed (Participants) | 106 | 98
units on a scale
  12 weeks | -2.2 [-3.7 to -0.9] | 0.5 [-1 to 2]
  24 weeks | -1.7 [-3.1 to -0.4] | 0.2 [-1.3 to 1.7]
  52 weeks | -1.1 [-2.7 to 0.5] | -0.003 [-1.6 to 1.6]

7. Secondary Outcome: Change in Arthritis Self-Efficacy Scale
Description: The Arthritis Self-Efficacy Scale is a self-report score measuring self-efficacy with respect to arthritis (range, 1 to 10, with higher scores indicating greater self-efficacy).
Time Frame: From Week 0, to Week 12, or to week 24, or to week 52
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi | Physical Therapy
Number analyzed (Participants) | 106 | 98
units on a scale
  12 weeks | 1.3 [0.8 to 1.8] | 0.8 [0.3 to 1.4]
  24 weeks | 0.9 [0.4 to 1.4] | 0.9 [0.4 to 1.4]
  52 weeks | 1.0 [0.5 to 1.5] | 0.7 [0.2 to 1.2]

8. Secondary Outcome: Change in Short-Form Health Survey (SF-36) Mental Component Score (MCS)
Description: The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) Mental Component Score (MCS) is the summary score for the mental quality-of-life components (range, 0 to 100, with higher scores indicating better health status)
Time Frame: From Week 0, to Week 12, or to week 24, or to week 52
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi | Physical Therapy
Number analyzed (Participants) | 106 | 98
units on a scale
  12 weeks | 1.6 [-0.1 to 3.2] | -0.03 [-1.7 to 1.7]
  24 weeks | 0.4 [-1.5 to 2.2] | -0.7 [-2.7 to 1.4]
  52 weeks | -0.1 [-1.9 to 1.8] | -1.5 [-3.4 to 0.4]

9. Secondary Outcome: Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Physical Function
Description: The WOMAC (version VA3.1) is a validated, self-administered, visual analogue scale specifically designed to evaluate knee and hip osteoarthritis. It has three subscales that are analyzed separately: pain (score range, 0-500), stiffness (0-200), and function (0-1700), with higher scores indicating more severe disease.
Time Frame: From Week 0, to Week 12, or to week 24, or to week 52
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi | Physical Therapy
Number analyzed (Participants) | 106 | 98
units on a scale
  12 weeks | -608.3 [-695.3 to -521.4] | -114.1 [-240 to 118]
  24 weeks | -586.8 [-669.5 to -504.1] | -455.7 [-543.1 to -368.4]
  52 weeks | -532.3 [-625.9 to -438.7] | -444.0 [-541.3 to -346.7]

10. Secondary Outcome: Outcome Expectation Scale
Description: The Outcome Expectations for Exercise Scale (range, 1 to 5, with 1 indicating no expectations for exercise and 5 the highest expectations for exercise) is a self-report measure of outcome expectations for exercise.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tai Chi | Physical Therapy
Number analyzed (Participants) | 106 | 98
units on a scale | 3.9 (0.5) | 3.9 (0.6)

11. Secondary Outcome: Change in Western Ontario and McMasters University Osteoarthritis Index (WOMAC) Pain Subscale
Description: as for outcome 9
Time Frame: From Week 0, to week 24 or to week 52
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi | Physical Therapy
Number analyzed (Participants) | 106 | 98
units on a scale
  24 weeks | -158.6 [-182.9 to -134.3] | -124.3 [-150.0 to -98.5]
  52 weeks | -138.8 [-166.7 to -110.8] | -121.0 [-150.0 to -91.9]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: participants are monitored weekly during intervention for adverse events. All are recorded on a case report form and evaluated according to Institutional Review Board mandated criteria. No systematic ascertainment of adverse events is undertaken after the intervention period based on the principle that all would be unrelated to the intervention.
Arm/Group | Tai Chi | Physical Therapy
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/98
Other Adverse Events (participants affected / at risk) | 0/106 | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No